CLINICAL TRIAL: NCT06943833
Title: A Phase II Single-arm Multi-centre Study of Volrustomig in Women With High Risk Locally Advanced Cervical Cancer Who Have Not Progressed Following Platinum Based, Concurrent Chemoradiation Therapy
Brief Title: A Study of Volrustomig in Women With High Risk Locally Advanced Cervical Cancer (IVOLGA)
Acronym: IVOLGA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZ-RU-00011
Record Dates: First submitted 2025-03-11; First posted 2025-04-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Cervical Cancer
Keywords: Locally Advanced Cervical Cancer;; Volrustomig

STUDY DESIGN:
Intervention Model Description: All participants will receive volrustomig as IV infusions
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Volrustomig
  Interventions: Biological: Volrustomig

INTERVENTIONS:
Biological: Volrustomig — IV infusion
  Other Names: MEDI5752

SUMMARY:
This is a phase II single-arm open-label study to investigate the efficacy and safety of volrustomig in women with FIGO 2018 stage IIIA to IVA cervical cancer who have not progressed following platinum-based concurrent chemoradiation therapy (CCRT).

DETAILED DESCRIPTION:
This is a phase II, single-arm open-label study to explore the efficacy and safety of volrustomig (MEDI5752) in women with high-risk locally advanced cervical cancer (Federation of Gynecologists and Obstetricians (FIGO) 2018 Stage IIIA to IVA) who have not progressed following platinum-based CCRT.

All participants will be assigned to receive volrustomig as intravenous (IV) infusions for up to end of treatment, or until Response Evaluation Criteria in Solid Tumors (RECIST) 1.1-defined radiological progression or histopathologically confirmed progression by Investigator assessment, unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met.

The results of this study will provide clinical data on efficacy and safety of an innovation treatment in the new region - Russian Federation.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, patients should fulfill the following criteria:

* Female.
* Aged at least 18 years at the time of screening.
* Body weight > 35 kg.
* Histologically documented FIGO 2018 Stage IIIA to IVA cervical adenocarcinoma, cervical squamous carcinoma, or cervical adenosquamous carcinoma, with no evidence of metastatic disease.
* Initial staging procedures performed no more than 42 days prior to the first dose of CCRT.
* Known PD-L1 status.
* Must not have progressed following CCRT.
* World Health Organization/The Eastern Cooperative Oncology Group (WHO/ECOG) performance status of 0 or 1.
* Adequate organ and bone marrow function.
* Capable of providing signed informed consent.

Exclusion Criteria:

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

* Diagnosis of small cell (neuroendocrine) or mucinous adenocarcinoma of cervical cancer.
* Evidence of metastatic disease.
* Intent to administer a fertility-sparing treatment regimen.
* History of organ transplant or allogenic stem cell transplant.
* Active or prior documented autoimmune or inflammatory disorders.
* Uncontrolled intercurrent illness.
* History of another primary malignancy except for a) Malignancy treated with curative intent with no known active disease ≥2 years before the first dose of study intervention; b) Adequately treated nonmelanoma skin cancer or lentigo maligna, or carcinoma in situ without evidence of disease.
* Unresolved toxicities from previous CCRT except for irreversible toxicity that is not reasonably expected to be exacerbated.
* Prior history or presence of vesicovaginal, colovaginal, or rectovaginal fistula.
* History of anaphylaxis to any biologic therapy or vaccine.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of the study intervention is excluded. The following are exceptions to this criterion: a) Intranasal, inhaled, topical steroids, or local steroid injections (eg, intraarticular injection); b) Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication or chemotherapy premedication) or a single dose for palliative purpose (eg, pain control).
* Patients who have undergone a previous hysterectomy, including a supracervical hysterectomy, or will have a hysterectomy as part of their initial cervical cancer therapy.
* Any prior (besides prior CCRT) or concurrent treatment for cervical cancer.
* Major surgical procedures within 4 weeks prior to the first dose of the study intervention or still recovering from prior surgery.
* Exposure to immune mediated therapy prior to the study for any indication.
* Receipt of live attenuated vaccine within 30 days prior to the first dose of the study intervention.
* Participants with a known allergy or hypersensitivity to the study intervention, or any excipients of the study intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 30 (Actual)
Dates: Start 2025-03-31 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival at 24 months (PFS24) | From date of first dose until 24 months.
  PFS24 is defined as the Kaplan-Meier estimate of PFS at 24 months per RECIST 1.1 or histopathologically confirmed progression as assessed by the Investigator or death due to any cause, whichever occurs earlier.

SECONDARY OUTCOMES:
Overall Survival at 36 months (OS36) | From date of first dose until 36 months.
  OS36 is defined as the Kaplan-Meier estimate of OS at 36 months after study drug administration.
Progression-free Survival at 36 months (PFS36) | From date of first dose until 36 months.
  PFS36 is defined as the Kaplan-Meier estimate of PFS at 36 months per RECIST 1.1- defined radiological progression or histopathologically confirmed progression as assessed by the Investigator or death due to any cause, whichever occurs earlier.
Time to First Subsequent Therapy or death (TFST) | From date of first dose until 36 months.
  TFST: The time from randomization until the start date of the first subsequent anti-cancer therapy after discontinuation of randomized treatment, or death due to any cause.

OTHER OUTCOMES:
Incidence of adverse events of Volrustomig | From the time of ICF signature up to 48 months.
  An adverse event is defined as the development of any untoward medical occurrence (other than progression of the malignancy under evaluation) in a patient or clinical study participant administered a medicinal product, and which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Locations (6):
- Russia (6):
  - Research Site, Arkhangelsk
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Ufa
  - Research Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/